CLINICAL TRIAL: NCT06349278
Title: Pancreatic Cancer and Synchronous Liver Metastases Resection Following Neoadjuvant FOLFIRINOX: a Prospective, Pilot Study
Brief Title: Pancreatic Cancer and Synchronous Liver Metastases Resection Following Neoadjuvant FOLFIRINOX
Acronym: PDAC-LIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alexandre Brind'Amour, Principal investigator, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-7276
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Adenocarcinoma; Pancreas Metastases; Pancreas Cancer
Keywords: PDAC; Liver metastases; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: One group will undergo intervention prospectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will undergo surgery for primary pancreatic cancer and liver metastases.
  Interventions: Procedure: Pancreatic resection and non-anatomic liver resections.

INTERVENTIONS:
Procedure: Pancreatic resection and non-anatomic liver resections. — Pancreatic resection and non-anatomic liver resections.

SUMMARY:
This is a prospective, pilot study from a single center. Patients will be evaluated and operated on by one of five surgeons with a subspeciality in hepato-biliary and pancreatic surgery. After thorough, standard of care assessment for both pancreatic primary and liver metastases resectability with blood tumor markers (CEA, CA 19-9 and CA-125), triphasic CT-scan and liver magnetic resonance imaging (MRI), patients with resectable pancreatic ductal adenocarcinoma primary and three or less resectable liver metastases will be prospectively included in the study. PET-scan may be added to the investigation depending on CT-scan or MRI results to prove metastatic disease or rule out extrahepatic metastases. Patients will receive a total of 12 cycles of perioperative FOLFIRINOX (FFX), with first reassessment with triphasic CT-scan to monitor tumor response after the first six cycles. Every patient will receive at least 6 cycles of FFX before surgery. The remaining six cycles will be received either preoperatively or postoperatively, depending on patient tolerance and tumor response at reassessment. Patients with liver metastases only visible on MRI will also have liver MRI at reassessment, which is also standard of care. Patients with evidence of tumor response on both imaging using RECIST V.1.1 criteria (stable disease or partial response), and blood tumor markers (≥ 80% decrease and/or normalization of all tumor markers) will then undergo pancreatic resection, either distal pancreatectomy or pancreatoduodenectomy depending on tumor side, with liver metastases excision. Each case will be followed with blood tumor markers and CT-scan every three months for two years, and every four months afterwards or until recurrence, which is standard of care for patients with metastatic PDAC. For patients without evidence of tumor response on imaging, or < 80% decrease of all tumor markers, the standard palliative systemic treatment will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pancreatic ductal adenocarcinoma (PDAC).
* Resectable primary tumor based on triphasic CT-scan.
* ≤ 3 liver metastases.
* Liver resections can be performed by local excision or non-anatomical, partial hepatectomy. Patients with complete radiologic response after neoadjuvant FOLFIRINOX (FFX), therefore not requiring liver resection, will be included.
* No evidence of extrahepatic metastases.
* Patient fit for pancreatic resection (ECOG 0 or 1).
* Stable or partial response on imaging after neoadjuvant FFX.
* No new metastasis after neoadjuvant FFX
* Blood tumor markers ≥ 80% decreased or within normal values after neoadjuvant FFX.

Exclusion Criteria:

* Impossibility to obtain tissue diagnosis preoperatively confirming PDAC.
* Locally advanced disease on triphasic CT-scan.
* > 3 liver metastases.
* Major hepatectomy required for liver metastases (right hepatectomy, left hepatectomy, central hepatectomy, extended right or left hepatectomy).
* Suspicion or confirmation of extrahepatic metastases.
* Patient unfit for pancreatic resection (ECOG 2 or more).
* Contraindication to receive FFX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2029-01-16 (Estimated)

PRIMARY OUTCOMES:
Morbidity and mortality | 90 days
  Post-operative complications

SECONDARY OUTCOMES:
Overall survival | 3 years after surgery
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Brind'Amour, MD, MSc, Principal Investigator — CHU de Québec
Locations (1):
- CHU de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD sharing.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] De La Cruz MS, Young AP, Ruffin MT. Diagnosis and management of pancreatic cancer. Am Fam Physician. 2014 Apr 15;89(8):626-32. PMID 24784121
- [Background] Rawla P, Sunkara T, Gaduputi V. Epidemiology of Pancreatic Cancer: Global Trends, Etiology and Risk Factors. World J Oncol. 2019 Feb;10(1):10-27. doi: 10.14740/wjon1166. Epub 2019 Feb 26. PMID 30834048
- [Background] Hishinuma S, Ogata Y, Tomikawa M, Ozawa I, Hirabayashi K, Igarashi S. Patterns of recurrence after curative resection of pancreatic cancer, based on autopsy findings. J Gastrointest Surg. 2006 Apr;10(4):511-8. doi: 10.1016/j.gassur.2005.09.016. PMID 16627216
- [Background] Sohal DPS, Kennedy EB, Khorana A, Copur MS, Crane CH, Garrido-Laguna I, Krishnamurthi S, Moravek C, O'Reilly EM, Philip PA, Ramanathan RK, Ruggiero JT, Shah MA, Urba S, Uronis HE, Lau MW, Laheru D. Metastatic Pancreatic Cancer: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2018 Aug 20;36(24):2545-2556. doi: 10.1200/JCO.2018.78.9636. Epub 2018 May 23. PMID 29791286
- [Background] Ducreux M, Cuhna AS, Caramella C, Hollebecque A, Burtin P, Goere D, Seufferlein T, Haustermans K, Van Laethem JL, Conroy T, Arnold D; ESMO Guidelines Committee. Cancer of the pancreas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v56-68. doi: 10.1093/annonc/mdv295. No abstract available. PMID 26314780
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Chun JW, Lee SH, Kim JS, Park N, Huh G, Cho IR, Paik WH, Ryu JK, Kim YT. Comparison between FOLFIRINOX and gemcitabine plus nab-paclitaxel including sequential treatment for metastatic pancreatic cancer: a propensity score matching approach. BMC Cancer. 2021 May 11;21(1):537. doi: 10.1186/s12885-021-08277-7. PMID 33975561
- [Background] Otsuka T, Shirakawa T, Shimokawa M, Koga F, Kawaguchi Y, Ueda Y, Nakazawa J, Komori A, Otsu S, Arima S, Fukahori M, Okabe Y, Makiyama A, Taguchi H, Honda T, Shibuki T, Nio K, Ide Y, Mizuta T, Mitsugi K, Ureshino N. A multicenter propensity score analysis of FOLFIRINOX vs gemcitabine plus nab-paclitaxel administered to patients with metastatic pancreatic cancer: results from the NAPOLEON study. Int J Clin Oncol. 2021 May;26(5):941-950. doi: 10.1007/s10147-021-01859-2. Epub 2021 Jan 23. PMID 33483857
- [Background] Lee JC, Woo SM, Shin DW, Kim J, Yang SY, Kim MJ, Kim JW, Kim JW, Lee WJ, Cha HS, Park P, Kim J, Hwang JH. Comparison of FOLFIRINOX and Gemcitabine Plus Nab-paclitaxel for Treatment of Metastatic Pancreatic Cancer: Using Korean Pancreatic Cancer (K-PaC) Registry. Am J Clin Oncol. 2020 Sep;43(9):654-659. doi: 10.1097/COC.0000000000000730. PMID 32889836
- [Background] Assenat E, de la Fouchardiere C, Portales F, Ychou M, Debourdeau A, Desseigne F, Iltache S, Fiess C, Mollevi C, Mazard T. Sequential first-line treatment with nab-paclitaxel/gemcitabine and FOLFIRINOX in metastatic pancreatic adenocarcinoma: GABRINOX phase Ib-II controlled clinical trial. ESMO Open. 2021 Dec;6(6):100318. doi: 10.1016/j.esmoop.2021.100318. Epub 2021 Nov 24. PMID 34837745
- [Background] Sakaguchi T, Valente R, Tanaka K, Satoi S, Del Chiaro M. Surgical treatment of metastatic pancreatic ductal adenocarcinoma: A review of current literature. Pancreatology. 2019 Jul;19(5):672-680. doi: 10.1016/j.pan.2019.05.466. Epub 2019 Jun 7. PMID 31285145
- [Background] Crippa S, Cirocchi R, Weiss MJ, Partelli S, Reni M, Wolfgang CL, Hackert T, Falconi M. A systematic review of surgical resection of liver-only synchronous metastases from pancreatic cancer in the era of multiagent chemotherapy. Updates Surg. 2020 Mar;72(1):39-45. doi: 10.1007/s13304-020-00710-z. Epub 2020 Jan 29. PMID 31997233
- [Background] Hashimoto D, Satoi S, Fujii T, Sho M, He J, Hackert T, Del Chiaro M, Jang JY, Gulla A, Yoon YS, Shan YS, Lou W, Valente R, Furuse J, Oba A, Nagai M, Terai T, Tanaka H, Sakai A, Yamamoto T, Yamaki S, Matsumoto I, Murakami Y, Takaori K, Takeyama Y. Is surgical resection justified for pancreatic ductal adenocarcinoma with distant abdominal organ metastasis? A position paper by experts in pancreatic surgery at the Joint Meeting of the International Association of Pancreatology (IAP) & the Japan Pancreas Society (JPS) 2022 in Kyoto. Pancreatology. 2023 Sep;23(6):682-688. doi: 10.1016/j.pan.2023.07.005. Epub 2023 Jul 20. PMID 37507301